CLINICAL TRIAL: NCT00307125
Title: B-Cell Depletion by Anti-CD20 (Rituximab) in Renal Allograft Recipients Who Develop Early De Novo Anti-HLA Alloantibodies Will Result in Inhibition of Alloantibody Production and Attenuation of Chronic Humoral Rejection
Brief Title: Rituximab in Renal Allograft Recipients Who Develop Early De Novo Anti-HLA Alloantibodies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network); Cooperative Clinical Trials in Pediatric Transplantation (CCTPT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-02; CCTPT-02 (Other: NIAID)
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Kidney Transplant; Kidney Transplant Recipient; Graft Function/Survival; de Novo HLA Antibodies Development
Keywords: Organ Transplantation; Graft function/survival; Immunosuppression; anti-CD20 (rituximab)
MeSH Terms: interventions — Rituximab; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilot Phase-Rituximab plus immunosuppression (Experimental): Enrollment into a Stage 2 pilot treatment study will occur after Stage 1. Adult Rituximab Dosing (Subjects > 18 years): 1000 mg on days 0 and 14; Pediatric Rituximab Dosing (Subjects <\=18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression is site-specific.
  Interventions: Drug: Rituximab plus immunosuppression
- Pilot Phase-Placebo plus immunosuppression (Placebo Comparator): Adult Placebo Dosing (Subjects >18 years): 1000 mg on days 0 and 14; Pediatric Placebo Dosing (Subject <\=18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression is site-specific.
  Interventions: Drug: Placebo plus immunosuppression

INTERVENTIONS:
Drug: Rituximab plus immunosuppression — Genetically engineered monoclonal antibody directed against the CD20 antigen on B cells and is known to deplete B cells when administered intravenously. Generally used in the treatment of non-Hodgkin's lymphoma
  Standard immunosuppression is site-specific.
  Other Names: Rituxan®; MabThera®; anti-CD20
  Arms: Pilot Phase-Rituximab plus immunosuppression
Drug: Placebo plus immunosuppression — Placebo dosing: Adult Dosing (Subjects >18 years): 1000 mg on days 0 and 14; Pediatric Dosing (Subject <\=18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression is site-specific.
  Other Names: Placebo for rituximab
  Arms: Pilot Phase-Placebo plus immunosuppression

SUMMARY:
The purpose of this study is to determine whether treatment with rituximab (anti-CD20, Rituxan®, MabThera®) in individuals who develop new anti-HLA antibodies after renal (kidney) transplant will promote longer-term survival of the transplanted kidney.The pilot study compares the use of rituximab (Rituxan®) + site-specific standard immunosuppression to placebo + site-specific standard immunosuppression in the treatment of circulating anti-HLA antibodies in subjects who develop de novo anti-HLA antibodies between 3-36 months after transplant.

DETAILED DESCRIPTION:
Organ rejection occurs when a patient's body does not recognize the new organ and attacks it. Data suggest that the development of anti-human leukocyte antigen (HLA) antibodies is an early clinical indication that organ rejection may occur. Rituximab is a genetically engineered monoclonal antibody directed against the CD20 antigen on B cells and is known to deplete B cells when administered intravenously; it is FDA-approved for the treatment of non-Hodgkin's lymphoma; Chronic Lymphocytic Leukemia (CLL); and Rheumatoid Arthritis (RA) in combination with methotrexate in adult patients with moderately-to severely-active RA who have inadequate response to one or more TNF antagonist therapies.

In a previous small study, kidney transplant patients with either acute humoral rejection (AHR) or chronic humoral rejection (CHR) were given rituximab and other antilymphocyte therapy. Patients with AHR had lower or undetectable levels of circulating anti-HLA antibodies after study treatment, and patients with CHR had a sustained decrease of anti-HLA antibodies to undetectable after 6 to 9 months.

This study will evaluate the safety and efficacy of rituximab in 1.)preventing organ rejection and 2.)promoting long-term survival of donor kidneys in people who undergo kidney transplantation.

This study involves two stages:

1. Stage 1 begins 3 to 36 months after transplant. During Stage 1, blood collection will occur every 3 months for up to 36 months after transplant to test for anti-HLA antibodies. When these antibodies are detected twice within 1 month, the patient will undergo a baseline kidney biopsy and have his or her glomerular filtration rate (GFR) measured to determine kidney function. If a patient meets certain study criteria, he or she will enter Stage 2 (Pilot Treatment Study).

   If anti-HLA antibodies are not detected in a patient's blood during Stage 1, the patient's participation will be complete.
2. In Stage 2, patients will receive site-specific standard immunosuppression plus randomization to either rituximab or placebo:

   * Adult dosing (>18 years of age), will receive an intravenous infusion of 1000mg of rituximab on Days 0 and 14.
   * Pediatric dosing (<\= than 18 years of age) will receive an intravenous infusion of 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses of rituximab on Days 0, 8, 15 and 22.

Adult participants will have 7-9 study visits over 12-24 months. Pediatric participants will have 9-11 study visits over 12-24 months. A physical exam, medication history, adverse events assessment, and blood and urine collection will occur at all visits. A biopsy of the kidney transplant will occur at Stage 2 entry and Month 12.

Note: Prior to January 2010, Stage 2 of this was a double-blind (double-masked) randomized pilot treatment study. As of January 2010 and beyond:

* subjects were no longer being recruited in the placebo treatment arm
* all treatment assignments were unblinded and an open-label design commenced; therefore, medication assignments were open to the study participants as well as to the site clinical team.
* all study subjects who participated in the study prior to this change were informed of the change
* all subjects who were randomized to the placebo-controlled arm and continued to meet the pilot study eligibility criteria were provided the option to participate in the pilot treatment study.

ELIGIBILITY:
Stage 1 Inclusion Criteria for All Participants:

* Willing to provide informed consent
* Previously diagnosed end stage renal disease (ESRD)
* Received kidney transplant within 3 and 36 months of study entry
* Willing to comply with the study protocol
* Willing to use acceptable forms of contraception during the study and for 12 months following rituximab/placebo therapy
* Willing to refrain from breastfeeding during the study and for 12 months following rituximab therapy

Stage 1 Inclusion Criteria for Pediatric Participants (<\=18 Years of Age):

* Parent or guardian willing to provide informed consent
* Have received all childhood vaccinations prior to study entry

Stage 2 Inclusion Criteria for Pilot Treatment Study:

* Three to 39 months post-transplant
* Developed new antibodies detected at two time points within 1 month between 3 to 36 months post-transplant
* Negative pregnancy test

Stage 1 Exclusion Criteria for All Participants:

* Recipient of a kidney from a donor older than 70 years of age
* Multi-organ transplant
* History of organ transplantation other than current kidney transplantation
* Previous treatment with rituximab
* History of severe allergic reactions to monoclonal antibodies
* History of allergic reaction to iodine glomerular filtration rate (GFR) assay
* Lack of intravenous (IV) access
* Sensitized to greater than 5% Panel Reactive Antibody (PRA) within 12 weeks prior to transplant
* History of recurrent bacterial or other significant infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis [TB] or atypical mycobacterial disease) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of study entry. Patients with fungal infections of nail beds are not excluded.
* HIV infected
* Surface antigen positive for hepatitis B virus (HBV)
* Antibody positive for hepatitis C virus (HCV)
* History of drug, alcohol, or chemical abuse within 6 months prior to study entry
* History of cancer. Patients with adequately treated in situ cervical carcinoma or adequately treated basal or squamous cell carcinoma of the skin are not excluded.
* Clinically significant cardiovascular or pulmonary disease
* Evidence of urinary tract obstruction causing decreased kidney function, unless corrected by study entry
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that would contraindicate use of an investigational drug, may affect interpretation of study results, or put the patient at high risk for treatment complications
* History of psychiatric disorder that may interfere with participation in the study
* History of nonadherence to prescribed regimens
* Use of other investigational drugs within 4 weeks of study entry
* Received any licensed or investigational live attenuated vaccine within 2 months of study entry.

Stage 2 Exclusion Criteria for All Participants:

* Previous treatment with rituximab
* Immunoglobulin Levels <500mg/dL (Combined IgM, IgG, IgA, IgE, IgD)
* History of severe allergic reactions to monoclonal antibodies
* History of cancer. Patients with adequately treated in situ cervical carcinoma or adequately treated basal or squamous cell carcinoma of the skin are not excluded.
* Active systemic infection at the time of entry into Stage 2
* Recurrent or de novo glomerular disease or Banff Grade III chronic rejection other than chronic humoral rejection (CHR) indicated in baseline kidney biopsy post-transplant
* History of post-transplant lymphoproliferative disease (PTLD)
* Serum creatinine of 3.0 mg/dl or greater OR GFR less than 25 ml/min at the time of entry into Stage 2
* Hemoglobin less than 8.5 g/dl
* Platelets less than 80,000 cells/mm^3
* White blood cell count less than 3,000 cells/mm^3
* AST or ALT 2.5 times the upper limit of normal at study entry
* Pregnant or breast-feeding
* Absolute neutrophil count less than 1000/mm^3

Stage 2 Exclusion Criteria for Pediatric Participants (<\=18 Years of Age):

* Positive test for parvovirus (B19) by PCR in the blood.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H. Sayegh, MD, Principal Investigator — Brigham and Women's Hospital; William Harmon, MD, Principal Investigator — Boston Children's Hospital; Anil Chandraker, MD, Study Chair — Brigham and Women's Hospital
Locations (17):
- United States (17):
  - University of Alabama, Pediatric Nephrology, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Illinois, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Legacy Transplant Services, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington

REFERENCES:
- [Background] Lee PC, Terasaki PI, Takemoto SK, Lee PH, Hung CJ, Chen YL, Tsai A, Lei HY. All chronic rejection failures of kidney transplants were preceded by the development of HLA antibodies. Transplantation. 2002 Oct 27;74(8):1192-4. doi: 10.1097/00007890-200210270-00025. PMID 12438971
- [Background] Mauiyyedi S, Colvin RB. Humoral rejection in kidney transplantation: new concepts in diagnosis and treatment. Curr Opin Nephrol Hypertens. 2002 Nov;11(6):609-18. doi: 10.1097/00041552-200211000-00007. PMID 12394606
- [Background] Worthington JE, Martin S, Al-Husseini DM, Dyer PA, Johnson RW. Posttransplantation production of donor HLA-specific antibodies as a predictor of renal transplant outcome. Transplantation. 2003 Apr 15;75(7):1034-40. doi: 10.1097/01.TP.0000055833.65192.3B. PMID 12698094
- [Derived] Fishman JA, Ikle DN, Wilkinson RA. Discrepant serological assays for Pneumococcus in renal transplant recipients - a prospective study. Transpl Int. 2017 Jul;30(7):689-694. doi: 10.1111/tri.12959. Epub 2017 May 2. PMID 28346714
- See also: Click here for the Clinical Trials in Organ Transplantation (CTOT) public Web site — http://www.ctotstudies.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N=757 subjects were enrolled in the screening phase (Stage 1: Screening) of the study and followed for development of de novo anti-HLA antibodies for up to 60 months post-kidney (renal) transplant.N=22 subjects from the screening cohort were enrolled in the treatment phase. Refer to Detailed Description and Eligibility Sections for more details.
Pre-assignment Details: From the screening cohort, N=22 subjects were enrolled in the treatment phase of the study (Stage 2: Pilot Study). Refer to Detailed Description and Eligibility Sections for more details.
Groups:
- Screening Phase: Kidney (renal) transplant recipients with no detectable anti-human leukocyte antigen (HLA) antibodies prior to transplant. Participants were screened for the development of anti-HLA antibodies once every 3 months up to 36 months post-transplantation and yearly thereafter until Month 60.
- Pilot Phase-Rituximab Plus Immunosuppression: Adult Dosing (Subjects > 18 years): 1000 mg on days 0 and 14; Pediatric Dosing (Subjects <\=18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression was site-specific.
- Pilot Phase-Placebo Plus Immunosuppression: Adult Dosing (Subjects >18 years): 1000 mg on days 0 and 14; Pediatric Dosing (Subject <\=18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression was site-specific.
Period: Screening Phase
Arm/Group | Screening Phase | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Started | 757 | 0 | 0
Completed | 303 | 0 | 0
Not Completed | 454 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 27 | 0 | 0
Not completed — Lost to Follow-up | 87 | 0 | 0
Not completed — Death | 10 | 0 | 0
Not completed — Withdrawal by Subject | 77 | 0 | 0
Not completed — Physician Decision | 26 | 0 | 0
Not completed — Sponsor Decision | 4 | 0 | 0
Not completed — Study Terminated | 17 | 0 | 0
Not completed — Graft Loss | 3 | 0 | 0
Not completed — Graft Failure | 8 | 0 | 0
Not completed — Follow-up period ended on Dec 31, 2011 | 83 | 0 | 0
Not completed — Scheduling issues/Non-compliance | 55 | 0 | 0
Not completed — Moved or transferred facilities | 34 | 0 | 0
Not completed — Received Pancreas Transplant | 8 | 0 | 0
Not completed — Ineligible for pilot | 4 | 0 | 0
Not completed — Try to get pregnant | 1 | 0 | 0
Not completed — Developed acute leukemia | 1 | 0 | 0
Not completed — Metastatic colon cancer | 1 | 0 | 0
Not completed — Malignancy | 1 | 0 | 0
Not completed — PAK | 1 | 0 | 0
Not completed — Ineligible | 1 | 0 | 0
Not completed — Screen Error | 1 | 0 | 0
Not completed — Sample of Anti-HLA Ab was not obtained | 1 | 0 | 0
Not completed — AMR and treated with rituximab | 1 | 0 | 0
Not completed — Coronary artery bypass | 1 | 0 | 0
Period: Pilot Phase
Arm/Group | Screening Phase | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Started | 0 | 15 | 7
Completed | 0 | 13 (2 participants had reduced follow-up) | 6 (1 participant had reduced follow-up)
Not Completed | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (19.5) | 49.0 (15.0) | 43.8 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: During Screening Phase: Incidence of Alloantibody Development
Description: Data were analyzed for 653 participants from the screening phase of the study. This outcome looked at the number of kidney transplant recipients that developed de novo HLA antibodies (anti-HLA Ab) post-transplant. Alloantibody is defined as an antibody produced following the introduction of an alloantigen into the system of an individual lacking that particular antigen. Alloantibodies are important mediators of acute and chronic rejection.
Time Frame: During screening window of 3-60 months post kidney transplant
Population: Screening sample
Measure: Number; unit: participants
Groups:
- Screening Phase: Participants who were analyzed during the screening phase/stage of the study
Arm/Group | Screening Phase
Number analyzed (Participants) | 653
participants | 79

2. Primary Outcome: During Screening Phase: Timing of Alloantibody Development
Description: Data were analyzed for 653 participants from the screening phase of the study. Of these, 79 (12%) developed de novo HLA-antibodies (anti-HLA Ab). This outcome looks at the average length of time (interval) from post kidney transplant until development of alloantibody. Alloantibody is defined as an antibody produced following the introduction of an alloantigen into the system of an individual lacking that particular antigen. Alloantibodies are important mediators of acute and chronic rejection
Time Frame: During screening window of 3-60 months post kidney transplant
Population: Screening sample
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Screening Phase: Participants who were analyzed during the screening phase of the study
Arm/Group | Screening Phase
Number analyzed (Participants) | 653
Months | 16.2 (9.9)

3. Primary Outcome: Number of Participants With 50 Percent (%) Decrease in Circulating Anti-Human Leukocyte Antigen (HLA) Antibodies
Description: Number of participants with 50% decrease in circulating anti-HLA antibodies at any time within the first 12 months post kidney transplant by LuminexTM Beads Method. Luminex assays for quantitation and detection of cytokine and signal transduction proteins. Presence of circulating antibodies is indicative of the transplant recipient's immune system responding to the transplanted organ as a foreign object or infection.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants | 2 | 0
Statistical Analysis 1: Comparison: Pilot Phase-Rituximab Plus Immunosuppression vs Pilot Phase-Placebo Plus Immunosuppression; Analysis by Fisher's exact test counting participants with 50% decrease in anti-HLA antibodies at any time within 12 months post treatment initiation; Test type: Superiority or Other; p > 0.999, Fisher Exact

4. Secondary Outcome: Number of Deaths 12 Months Post Treatment Initiation
Description: Number of participant deaths within 12 months post treatment initiation
Time Frame: 12 months post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Graft Loss 12 Months Post Treatment Initiation
Description: Number of participants with graft loss, defined as the need for dialysis for greater than 30 days duration, allograft nephrectomy, or the decision to withdraw immunosuppression due to graft failure within 12 month post treatment initiation
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Groups:
- Rituximab Plus Immunosuppression: Adult Dosing (Subjects > 18 years): 1000 mg on days 0 and 14; Pediatric Dosing (Subjects ≤18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression was site-specific.
- Placebo Plus Immunosuppression: Adult Dosing (Subjects >18 years): 1000 mg on days 0 and 14; Pediatric Dosing (Subject ≤18 years): 375 mg/m^2/dose (maximum 500 mg/dose) in 4 doses, once per week (Days 0, 8, 15 and 22).
  Standard immunosuppression is site-specific.
Arm/Group | Rituximab Plus Immunosuppression | Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Biopsy-proven Post-Transplant Lymphoproliferative Disease (PTLD)
Description: Number of participants with PTLD within 12 month post treatment initiation. Diagnosis of PTLD was made by B cell proliferation after therapeutic immunosuppression.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Loss of Peritubular Capillary (PTC) C4d Staining on Kidney Biopsy
Description: Number of participants with loss of PTC C4d staining on kidney (renal) biopsy within 12 months post treatment initiation. PTC C4d staining on biopsy indicates organ rejection.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants | 0 | 0

8. Secondary Outcome: Number of Participants With Viral Replication of Cytomegalovirus (CMV)
Description: Number of participants with viral replication of CMV within 12 month post treatment initiation. Measured by polymerase chain reaction (PCR) method. Evidence of viral replication is indicative of active CMV infection.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants
  Positive | 3 | 2
  Negative | 12 | 5
Statistical Analysis 1: Comparison: Pilot Phase-Rituximab Plus Immunosuppression vs Pilot Phase-Placebo Plus Immunosuppression; Test type: Superiority or Other; p > 0.999, Fisher Exact

9. Secondary Outcome: Number of Participants With Evidence of Viral Replication of Epstein-Barr Virus (EBV)
Description: Number of participants with positive viral replication of EBV within 12 month post treatment initiation. Measured by polymerase chain reaction (PCR) method. Evidence of EBV viral replication is indicative of active infection.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants
  Positive | 7 | 3
  Negative | 8 | 4
Statistical Analysis 1: Comparison: Pilot Phase-Rituximab Plus Immunosuppression vs Pilot Phase-Placebo Plus Immunosuppression; Test type: Superiority or Other; p > 0.999, Fisher Exact

10. Secondary Outcome: Number of Participants With Viral Replication of Polyomavirus (BKV)
Description: Number of participants with viral replication of BKV within 12 month post treatment initiation. Measured by polymerase chain reaction (PCR) method. Evidence of viral replication is indicative of a BKV infection. Polyomavirus BK is a significant pathogen in transplant recipients.
Time Frame: 1 year post treatment initiation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Number analyzed (Participants) | 15 | 7
participants
  Positive | 0 | 0
  Negative | 15 | 7

ADVERSE EVENTS:
Time Frame: From kidney (renal) transplant to the end of study
Description: Adverse events methods:
  * Observing the participant
  * Questioning the participant, which should be done in an objective manner.
  * Receiving an unsolicited complaint from the participant.
  * An abnormal value or result from a clinical or laboratory evaluation.
Arm/Group | Pilot Phase-Rituximab Plus Immunosuppression | Pilot Phase-Placebo Plus Immunosuppression
Serious Adverse Events (participants affected / at risk) | 5/15 | 1/7
Other Adverse Events (participants affected / at risk) | 3/15 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase-Rituximab Plus Immunosuppression (N=15) | Pilot Phase-Placebo Plus Immunosuppression (N=7)
Duodenal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Chlamydial pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase-Rituximab Plus Immunosuppression (N=15) | Pilot Phase-Placebo Plus Immunosuppression (N=7)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Slow accrual. In order to ensure the study was completed within the time frame allotted, randomization to the control arm (Pilot Phase-Placebo plus immunosuppression) was suspended. Enrollment continued to lag. The study was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No